CLINICAL TRIAL: NCT00713596
Title: The Use of Fibrin Sealant During Septorhinoplasty: Short and Long Term Benefits
Brief Title: Study Evaluating Benefit of Using Fibrin Glue in Septorhinoplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lead investigator moved to a new medical center; study was stopped when he left.
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-009614
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Results first posted 2012-07-24 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-03

CONDITIONS: Recovery Time; Bruising
Keywords: Nasal Surgery; Septorhinoplasty; fibrin glue; fibrinogen; Swelling; fibrin; tisseel
MeSH Terms: conditions — Contusions | interventions — Fibrinogen; Fibrin Tissue Adhesive; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (Sham Comparator): Septorhinoplasty with postoperative application of nasal taping and an external nasal cast. The tape and cast will be left in place for one week. No tissue glue will be used during the operation, although the nurse and surgical assistant will simulate the preparation and insertion of tissue glue using a syringe containing saline.
  Interventions: Procedure: Septorhinoplasty; Procedure: Taping after septorhinoplasty.; Procedure: Cast applied to the nose after nasal surgery; Other: Saline
- Fibrinogen, tape, and cast (Experimental): Septorhinoplasty will be performed. At the termination of the procedure, prior to closure, fibrin sealant will be applied by the surgical assistant to the surgical site. Approximately 0.5 cc to 2 cc of tissue sealant will be applied. After closure, tape and cast will be applied and left in place for one week.
  Interventions: Drug: Fibrinogen; Procedure: Septorhinoplasty; Procedure: Taping after septorhinoplasty.; Procedure: Cast applied to the nose after nasal surgery
- Fibrinogen and tape (Experimental): Septorhinoplasty will be performed. At the termination of the procedure, prior to closure, 0.5 cc to 2 cc of tissue sealant will be applied. Nasal tape will be applied after closure.
  Interventions: Drug: Fibrinogen; Procedure: Septorhinoplasty; Procedure: Taping after septorhinoplasty.

INTERVENTIONS:
Drug: Fibrinogen — One time application of 0.5 cc to 2.0 cc of fibrinogen following surgery.
  Other Names: Tisseel
  Arms: Fibrinogen and tape; Fibrinogen, tape, and cast
Procedure: Septorhinoplasty — Septorhinoplasty to correct nasal deviation.
Procedure: Taping after septorhinoplasty. — Simple taping over the nose following nasal surgery.
Procedure: Cast applied to the nose after nasal surgery — A molded cast will be placed on top of the nose following nasal surgery.
  Arms: Control group; Fibrinogen, tape, and cast
Other: Saline — Approximately 0.5 cc to 2 cc normal saline will be applied after the operation before the nasal taping and casting.
  Arms: Control group

SUMMARY:
The purpose of this study is to determine whether the use of fibrin glue during nasal surgery leads to a shorter recovery period with less bruising and/or swelling.

DETAILED DESCRIPTION:
Septorhinoplasty is a well established technique to correct nasal deformity. Drawbacks of this procedure include a significant recovery following surgery which may often require nasal taping and casting. Swelling and bruising in and around the surgical site may persist for months after the operation. At present, there is no standard regarding the length of time nasal tape and cast should be used following septorhinoplasty. It has never been proven that taping or casting is required - in surgeries that require minimal amounts of tissue handling, we may not use any tape or cast following the procedure. Homologous fibrin glue has been used for various cosmetic facial plastic procedures since the early 1980's. It has been shown to decrease bruising and swelling following surgery. This study is being undertaken to evaluate these benefits of using fibrin glue in nasal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Any patient over 18 years of age undergoing septorhinoplasty.

Exclusion Criteria:

* Any patient having more than one procedure performed during one anesthetic.(i.e.brow lift, face lift, blepharoplasty)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oren Friedman, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients presenting for septorhinoplasty at the Mayo Clinic, Rochester, MN were offered the opportunity to participate in the study.
Groups:
- Fibrin Sealant Group, Tape and Cast: Septorhinoplasty will be performed. At the termination of the procedure, prior to closure, fibrin sealant will be applied by the surgical assistant to the surgical site. Approximately 0.5 cc to 2 cc of tissue sealant will be applied. After closure, tape and cast will be applied and left in place for one week.
- Fibrin Sealant Group: Septorhinoplasty will be performed. At the termination of the procedure, prior to closure, 0.5 cc to 2 cc of tissue sealant will be applied. Nasal tape will be applied after closure.
Period: Overall Study
Arm/Group | Control Group | Fibrin Sealant Group, Tape and Cast | Fibrin Sealant Group
Started | 9 | 8 | 8
Completed | 7 | 5 | 6
Not Completed | 2 | 3 | 2
Not completed — Study was terminated | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Fibrin Sealant Group, Tape and Cast | Fibrin Sealant Group | Total
Number analyzed (Participants) | 9 | 8 | 8 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 8 | 25
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 10
  Male | 5 | 5 | 5 | 15
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 8 | 25

OUTCOME MEASURES:

1. Secondary Outcome: Assessment of the Results of Surgery 6 Months Post Operative by Review of Post Operative Photographs by the Operating Surgeon and 3 Blinded Reviewers Using a Mayo Clinic Surgeon Septorhinoplasty Questionnaire
Description: At the end of the study standard post operative rhinoplasty photos will be obtained, and the photos will be reviewed by three blinded observers, who are experienced rhinoplasty surgeons. The photos will be presented to the evaluators in a completely random fashion at a single session. These photos will be graded at that time using the same questionnaire used by the operating surgeon. The questionnaire covers bruising, swelling, tenderness, and length, width, hump and tip of nose, with a range 4-40, 4=ideal nose to 40=many postoperative problems and disfigured nose.
Time Frame: 6 months postoperative
Arm/Group | Control Group | Fibrin Sealant Group, Tape and Cast | Fibrin Sealant Group
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Patient Assessments of Disease-specific Quality of Life, Nasal Symptoms, and Nasal Form at 6 Months as Measured by Rhinoplasty Outcomes Evaluation (ROE), Nasal Obstructive Symptoms Evaluate Scale (NOSE), and Global Measure of Nose Deformity
Description: ROE: 6 items for subject's opinion re: nasal appearance, each item on 0-4 scale. Total score sum of 6 items, dividing total by 24 X 100, core ranges from 0 (least satisfied) to 100 (most satisfied).
  NOSE: Assess five conditions over the past month, each item on 0-4 scale X 5, then summed. Total score ranges from 0 (no problem) to 100 (severe problem).
  Global measure of nose deformity: Pictures of 4 indices of nasal anatomy: length, width, tip, and hump. Each index cored from 1-7, with 1=ideal nose, and 7=deformed nose. Total score = sum of 4 indices, range 4-28, lower score=more ideal nose
Time Frame: 6 months post operative
Arm/Group | Control Group | Fibrin Sealant Group, Tape and Cast | Fibrin Sealant Group
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Control Group | Fibrin Sealant Group, Tape and Cast | Fibrin Sealant Group
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Study was terminated due to principal investigator leaving the institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No